CLINICAL TRIAL: NCT01835691
Title: Differential Effects of Ergocalciferol and Cholecalciferol Therapies in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Jason Stubbs, MD, Assistant Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12861
Record Dates: First submitted 2013-04-12; First posted 2013-04-19 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Vitamin D; Vitamin D2; Vitamin D3
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D2 (ergocalciferol) (Experimental): 50,000 units once a week for 12 weeks
  Interventions: Dietary Supplement: Vitamin D2 (ergocalciferol)
- Vitamin D3 (cholecalciferol) (Experimental): 50,000 units once a week for 12 weeks
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)

INTERVENTIONS:
Dietary Supplement: Vitamin D2 (ergocalciferol) — 50,000 units once a week for 12 weeks
  Arms: Vitamin D2 (ergocalciferol)
Dietary Supplement: Vitamin D3 (cholecalciferol) — 50,000 units once a week for 12 weeks
  Arms: Vitamin D3 (cholecalciferol)

SUMMARY:
This study is to research two questions. First, is vitamin D3 more effective than vitamin D2 in raising 25-hydroxyvitamin D [25(OH)D] levels in chronic kidney disease (CKD) patients? And secondly, what are the differential effects of vitamin D2 and vitamin D3 on other mineral metabolism parameters?

DETAILED DESCRIPTION:
Vitamin D helps form and strengthens bones by allowing the body to absorb calcium. Vitamin D helps the immune system fight infection as well as helps keep muscles strong. Without enough vitamin D, bones can become weak, thin and brittle.

Vitamin D is useful in people with various types of health issues. Patients with CKD exhibit an unusually high rate of vitamin D deficiency, which may contribute to some of the poor clinical outcomes in this group.

This study will randomize patients with CKD and low vitamin D levels to two groups; one group will be treated with vitamin D2 (ergocalciferol) and the other group will be treated with vitamin D3 (cholecalciferol). The purpose of this study is to compare the effects of the two different forms of vitamin D specifically in patients chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Chronic kidney disease with an estimated glomerular filtration rate (GFR) between 15-60 ml/min (CKD stage III-IV)
* Vitamin D insufficiency (25-hydroxyvitamin D level < 30 ng/mL) that has not been treated with vitamin D replacement since the acquisition of this level

Exclusion Criteria:

* Current treatment with cholestyramine
* Presence of GI disorders such as short bowel, history of gastrectomy, colectomy, gastric bypass, inflammatory bowel disease, celiac disease, disorders of fat absorption, chronic diarrhea.
* Liver cirrhosis
* Known current substance abuse
* Current treatment with immunosuppressant medications
* Presence of chronic infection
* History of chronic inflammatory disease (i.e. - lupus, active rheumatoid arthritis, Crohns disease)
* Currently receiving high-dose vitamin D replacement (avg dose of ≥ 3,000 U per day) or "active" vitamin D analogue (e.g., calcitriol, which is 1,25-dihydroxyvitamin vitamin D).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in total serum 25-hydroxyvitamin D [25(OH)D] levels (ng/mL) | Baseline to immediately post-therapy (week 12)

SECONDARY OUTCOMES:
Change in serum 25-hydroxyvitamin D2 and D3 subfractions (ng/mL) | Baseline to immediately post-therapy (week 12), and week 12 to week 18
Change in total serum 25(OH)D (ng/mL) | week 12 to week 18
Change in serum intact parathyroid hormone (PTH) (pg/mL) | Baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Jason Stubbs, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States